CLINICAL TRIAL: NCT03902340
Title: Multicentre, Phase 3, Prospective Study With On-line Randomization, in Single Blind Conditions for the Primary Efficacy Endpoint, Controlled, in Two Parallel Groups, Comparing the Efficacy, Tolerability and Safety of actiTENS Versus Level 2 Systemic Analgesics Recommended for the Treatment of Chronic Nociceptive Pain of Moderate to Severe Intensity in Patients Suffering From Osteoarthritis of the Knee
Brief Title: Comparison of the Efficacy, Tolerability and Safety of actiTENS to Those of Level 2 Analgesic Treatments.
Acronym: ArthroTENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sublimed (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A01895-50
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
Keywords: Pain; Knee osteoarthritis (KOA); Nociceptive pain; TENS; Step 2 analgesics
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Nociceptive Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): Treatment by non-pharmacological transcutaneous electric nerve stimulation (TENS)
  Interventions: Device: ActiTENS
- level 2 systemic analgesic treatments (Active Comparator): Treatment by level 2 analgesic pharmacological treatment indicated in the treatment of chronic nociceptive pain of moderate to severe intensity.
  Interventions: Drug: Level 2 Analgesic Treatments

INTERVENTIONS:
Device: ActiTENS — ActiTENS is a rechargeable box, weighing 64g attached by Velcro to an adhesive support, which can be positioned on the skin at any position chosen by the patient. The patient will use the programme (P4) prescribed by his doctor and will regulate the intensity of stimulation using an application downloaded to his smartphone which will communicate with the box via Bluetooth.
  Arms: TENS
Drug: Level 2 Analgesic Treatments — There are 4 level 2 oral analgesic treatments indicated for chronic nociceptive pain of moderate to severe intensity (between 4 and 7 on a simple numerical scale of 11 points) (12):
  * Tramadol immediate release formulation (IR, one intake every 6 hours) or prolonged release formulation (PR, one intake every 12 hours); maximum posology 400mg/24h.
  * Dihydrocodeine: 60mg every 12 hours; maximum posology 120mg/24h.
  * Combination of paracetamol and codeine in a fixed combination every 6 hours; maximum posology of codeine: 300mg/24h.
  * Combination of paracetamol and tramadol in a fixed combination; maximum posology of tramadol: 8 tablets/24h ie 300mg/24h.
  Arms: level 2 systemic analgesic treatments

SUMMARY:
This is a phase 3, multicentre, prospective, single-blind on principal efficacy criterion, 2 parallel groups, randomized, controlled clinical study comparing efficacy and safety of actiTENS versus systemic level 2 analgesics recommended for the treatment of moderate or severe, nociceptive, chronic pain in patients suffering from osteoarthritis of the knee.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a debilitating chronic condition requiring long-term treatment of pain and inducing functional impairment. More specifically knee osteoarthritis (KOA) is a common disease associated with significant morbidity. Its prevalence increases with age dramatically. KOA is frequently associated with pain which can worsen with daily activities. The goals of KOA treatments are to provide pain relief and to improve function and quality of life. For the American college of Rheumatology and despite the frequent use of TENS in treating patients with KOA, questions remained regarding its efficacy. Consequently TENS needs additional clinical studies to demonstrate its efficacy in management of painful osteoarthritis.

The main objective of this study is to demonstrate the efficacy and to the safety of TENS in the management of chronic, nociceptive pain in patient suffering from KOA.

ELIGIBILITY:
Inclusion Criteria:

* Adult > or = 55 years.
* Being monitored by a rheumatologist in private practice or in a hospital.
* Presenting nociceptive pain:

  * chronic (for at least 3 months),
  * secondary to knee osteoarthritis confirmed by x-ray: stage 2 and over according to Kellgren and Lawrence.
* Of moderate to severe intensity equal to or above 4 on a numerical scale of 0-10.
* In a situation of analgesic therapy failure for level 1 analgesics:

  * paracetamol and NSAIDS,
  * Prescribed at therapeutic dose : 4 g/d of paracetamol and 1200 mg/d of ibuprofen or equivalent (analgesic dose),
  * For at least 2 weeks,
* Requiring a level 2 prescription.
* Affiliated to social security insurance.
* Informed of the concept and agreeing to use the TENS as a non-medicinal analgesic treatment.
* Capable of understanding how to use the TENS and the level 2 analgesic treatments.
* Intellectually and physically able to participate in the study in the opinion of the investigator.
* Owns a Smartphone to be able to download the actiTENS application.

Exclusion Criteria:

* Current or previous allergy to the actiTENS electrodes.
* On-going or planned pregnancy and absence of effective contraception (except for menopausal women).
* Neuropathic pain with a DN4 result > 4/10 or with a positive response to one or more questions in the DN4 clinical examination.
* Osteoarthritis flare.
* Surgery planned in the following 6 months.
* History of multiple operations on the knee concerned.
* Medicinal or non-medicinal treatments which could influence the pathology being studied.
* Modification of medicinal or non-medicinal treatments planned in the following 6 months.
* Current participation in another study.
* Presence of another painful condition which could perturb the evaluation.
* Patient with an absolute contraindication to TENS or level 2 systemic analgesic treatments recommended for the treatment of chronic pain of moderate or severe intensity.
* Patient unable to express his/her consent or deprived of liberty.
* Patient with cognitive disorder or behaviour rendering him/her unsuitable to follow the instructions for this study.
* Patient not affiliated to a social security system.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy : pain intensity evaluated by a numerus scale from 0 to 10 | 3 months after dosing
  Pain intensity (PI) at M3 between both treatment groups. Numerus scale with a minimum of 0 (no pain) to a maximum of 10 (maximum pain).
Safety : occurence of adverse events | 3 months after dosing
  Number of adverse events (AE) occurred during the 3 months of follow-up and due to studied treatments.

SECONDARY OUTCOMES:
Efficacy : pain intensity evaluated by a numerus scale from 0 to 10 | 1, 3 and 6 months after dosing
  Minimum, maximum,median and difference of pain intensity (PI) during movement and at rest at M1, M3 and M6 between both treatment groups
Efficacy : functional status evaluated by the WOMAC score (Western Onatario McMaster score) | 1, 3 and 6 months after dosing
  Functional status (pain, function, stiffness) at M1, M3 and M6.
Efficacy : pain relief (PAR) evaluated by the pain visual analogue scale (VAS) | 1, 3 and 6 months after dosing
  Pain relief at M1, M3 and M6. VAS from 0 to 10 with 0 = no relief and 10 = total relief). Scale of 100 mm.
Efficacy : quality of life evaluated by the questionnaire EuroQol-5D | 1, 3 and 6 months after dosing
  Evaluation of the quality of life at M1, M3 and M6
Efficacy : patient global impression of change evaluated by a global impression questionnaire. | 1, 3 and 6 months after dosing
  Evaluation of the change on activity, symptoms, emotions, quality of life regarding the pain of patient at M1, M3 and M6
Efficacy : drop-outs for inefficacy | Through study completion, an average of 6 months
  Evaluation of the number of patient drop outs because of treatment inefficacy in each arm
Efficacy : prolongation of studied treatment | Through study completion, an average of 6 months
  Evaluation of the number of patient wishes to continue the studied treatment.
Safety : occurrence of Adverse Events (AE) | Through study completion, an average of 6 months
  Evaluation by the type of AE and the date of occurence
Safety : drop-outs for AE and corrective treatments | Through study completion, an average of 6 months
  Evaluation of the number of patient drop outs because of the occurence of adverse events in each arm
Estimation of direct costs. | Through study completion, an average of 6 months
  Comparison of treatment costs between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CORTET, Pr, Principal Investigator — Hôpital Roger Salengro - Service de Rhumatologie
Locations (1):
- Hôpital Roger Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maheu E, Soriot-Thomas S, Noel E, Ganry H, Lespessailles E, Cortet B. Wearable transcutaneous electrical nerve stimulation (actiTENS(R)) is effective and safe for the treatment of knee osteoarthritis pain: a randomized controlled trial versus weak opioids. Ther Adv Musculoskelet Dis. 2022 Jan 18;14:1759720X211066233. doi: 10.1177/1759720X211066233. eCollection 2022. PMID 35069809